CLINICAL TRIAL: NCT00760604
Title: A Phase III Study of En Bloc Versus Non-En Bloc Esophagectomy in Patients With Locally Advanced Esophageal Cancer
Brief Title: A Phase III Study of En Bloc Versus Non-En Bloc Esophagectomy in Esophageal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed due to slow patient accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Paul C. Lee, Associate Professor of Cardiothoracic Surgery, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0806009855
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal neoplasms; Esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): En bloc esophagectomy is performed through a transthoracic approach by removing the tumor-bearing esophagus, the pericardium anteriorly, both pleural surfaces laterally, as well as the thoracic duct and all other lymphoareolar tissue wedged posteriorly between the esophagus and the spine, and en-bloc resection of all nodal groups in the middle and lower mediastinum as well as the upper abdomen.
  Interventions: Procedure: Esophagectomy
- B (Active Comparator): Transhiatal esophagectomy is performed through an abdominal incision and a neck incision. The stomach is mobilized, and the left gastric vessels are transected at its origin. Celiac lymph nodes are dissected, and the intrathoracic esophagus is dissected bluntly through the hiatus and through the neck. The cervical esophagus is divided at the level of the neck. After the esophagogastrectomy is performed, a gastric tube is created. An esophagogastrostomy is then performed in the neck. If a transthoracic approach is used, dissection will be as described for the transhiatal approach.
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — Comparison of en-bloc vs. non-en bloc esophagectomy

SUMMARY:
The purpose of this study is to test 2 different methods of surgery to remove cancer in the esophagus. This research is being done to see whether removing more tissue and lymph nodes surrounding the tumor in the esophagus (known as transthoracic en bloc esophagectomy) offers better control of the cancer than removing less tissue and lymph nodes (known as non-en bloc esophagectomy).

DETAILED DESCRIPTION:
The aim of this study is to determine the 5-year disease-free survival, overall survival, and time to progression comparing (Arm A) transthoracic en bloc esophagectomy and (Arm B) transhiatal or transthoracic non-en bloc esophagectomy. Randomization to the two surgical arms will take place after the patient has given written informed consent and eligibility has been established. Patients will be informed of their randomized arm prior to the day of surgery. Preoperative chemotherapy may be administered at the discretion of the treating physician. Adjuvant chemotherapy and/or radiotherapy will be prescribed at the discretion of the treating physician. All patients will be followed for recurrence and survival for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cT2-T3/N0-N1-M1a-M1b(lymph node metastasis only) esophageal squamous cell and adenocarcinoma who have potentially resectable disease.
* Karnofsky performance status greater than or equal to 80%.
* Pulmonary and cardiac function must be acceptable for surgery according to institutional standards.
* Acceptable hepatic, renal and bone marrow function.
* Age 18 or older.
* Patients may receive preoperative chemotherapy and/or radiation therapy as part of their clinical care.

Exclusion Criteria:

* Patients with clearly unresectable or metastatic esophageal cancer or clinical stage I esophageal cancer.
* Significant psychiatric illness that would interfere with patient compliance.
* Patients with any other serious underlying medical condition that would impair the ability of the patient to receive or comply with protocol treatment.
* Patients with a significant history of unstable cardiovascular disease (e.g., inadequately controlled hypertension, or angina; myocardial infarction within the previous 6 months; ventricular cardiac arrhythmias requiring medication; congestive heart failure that in the opinion of the treating physician should preclude the patient from protocol treatment.
* Uncontrolled diabetes mellitus or uncontrolled infection, including HIV or interstitial pneumonia or interstitial fibrosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Disease free survival defined as the time from surgical resection to the time of recurrent disease, death from esophageal cancer, or death from any cause. | CT scans will be performed every 6 months for 5 years.

SECONDARY OUTCOMES:
To determine 5-year overall and disease-specific survival in arm A and arm B | CT scans every 6 months for 5 years
To determine the rates of local and systemic recurrence in arm A vs. arm B | CT scans performed every 6 months for 5 years
To determine time to progression in arm A vs. arm B | CT scans every 6 months for 5 years
To determine mortality and morbidity in arm A vs. arm B | 5 years from the date of surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Lee, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell Unversity, New York, New York, United States